CLINICAL TRIAL: NCT04417075
Title: Culturally Sensitive, Evidence-based, Spanish Language Mobile App for Smoking Cessation for Latino Cigarette Smokers
Brief Title: Mobile Smoking Treatment for Spanish-speaking Latinx Smokers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Michael J. Zvolensky, Ph.D., Hugh Roy and Lillie Cranz Cullen Distinguished University Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001567; 1R41DA048692-01 (NIH)
Record Dates: First submitted 2020-05-30; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; Mobile App; Anxiety Sensitivity
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Impacto (Experimental): This is the mobile app to be developed and evaluated in this project.
  Interventions: Behavioral: Impacto (Mobile App)
- Dejar de Fumar Asistente (Active Comparator): This is the mobile app that will serve as the control condition in evaluating the efficacy of Impacto.
  Interventions: Behavioral: Dejar de Fumar Asistente (Mobile App)

INTERVENTIONS:
Behavioral: Impacto (Mobile App) — This is the mobile app to be developed and evaluated in this project. It is designed for Spanish-speaking, Latinx smokers with high anxiety sensitivity and will be built for the Android platform. The app will include components to address and remediate anxiety sensitivity, as well as having smoking cessation components.
  Arms: Impacto
Behavioral: Dejar de Fumar Asistente (Mobile App) — Dejar de Fumar Asistente (English version called: Quit Tracker: Stop Smoking) is a popular, free third party mobile application aimed at helping smokers quit smoking. This is the mobile app that will serve as the control condition in evaluating the efficacy of Impacto. This mobile app is well established as a smoking cessation app for Spanish-speaking, Latinx smokers. The app includes smoking cessation components but does not have a specific emphasis on anxiety sensitivity.
  Arms: Dejar de Fumar Asistente

SUMMARY:
The specific aims of the project are to develop and test a Spanish language, mobile app for smoking cessation called Impacto.

DETAILED DESCRIPTION:
A total of 38 Spanish-speaking, Latinx smokers with high anxiety sensitivity (AS) will be recruited for this project. Eight (8) participants will complete user interviews in Spanish and thirty (30) participants will participate in a randomized controlled trial (RCT) for smoking cessation. Participants will be randomized to receive either the Impacto mobile app or a generic, Spanish language, smoking cessation, mobile app control (Dejar de Fumar Asistente).

ELIGIBILITY:
Inclusion Criteria:

1) 18 to 55 year of age, 2) current smoker (i.e., at least 6 cigarettes/day), 3) not currently engaged in smoking cessation treatment, 4), high anxiety sensitivity (AS) score defined as an ASI-III score of ≥ 23, 5) motivation to quit > 5 on a 10 pt. scale, 6) Spanish speaking, and 7) currently own an Android-compatible mobile phone.

Exclusion Criteria:

1) use of other tobacco products (including e-cigarettes), 2) current non-nicotine substance dependence and/or current or intended participation in a concurrent substance abuse treatment, 3) ongoing psychotherapy of any duration directed specifically toward the treatment of anxiety or depression, or 4) active suicidality (i.e., suicidal ideation, intent, and/or plan) or current psychosis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-02-21 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
7-Day Point Prevalence Smoking Abstinence | End of treatment (Week 8)
  Self-reported 7-day point prevalence smoking status. Verification via carbon monoxide at end of treatment (10 weeks).
Change in Smoking Rate (# cigarettes per day) | Baseline and Weeks 2, 4, 6, and end of treatment (Week 8)
  We will assess the number of cigarettes smoking at each time point.

SECONDARY OUTCOMES:
Change in Anxiety Sensitivity | Baseline and Weeks 2, 4, 6, and end of treatment (Week 8)
  Anxiety sensitivity will be assessed using the Anxiety Sensitivity Index-3 (ASI-3).
Change in Mood and Anxiety Symptoms | Baseline and Weeks 2, 4, 6, and end of treatment (Week 8)
  The Mood and Anxiety Symptom Questionnaire (MASQ) is well-validated measure and will be used to assess anxiety/depressive symptoms.
Daily Adherence to Use of Impacto Mobile App (Impacto Condition Only) | Daily over the course of the 8 weeks of participant study involvement
  We will access these data via the "back end" of the Impacto server to evaluate whether the criterion of 75% daily adherence (i.e., app use on 75% of all possible days) has been achieved.
User Satisfaction with the Impacto Mobile App (Impacto Condition Only) Condition Only) | Weeks 2, 4, 6, and 8
  User satisfaction ratings scored on a 1-9 Likert scale with higher scores indicating better user satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Anxiety and Health Research Laboratory and Substance Use Treatment Clinic, University of Houston, Houston, Texas, United States